CLINICAL TRIAL: NCT00005059
Title: A Phase II Study of Carboplatin and Paclitaxel in Elderly Patients With Metastatic or Recurrent Unresectable Non-Small Cell Lung Cancer
Brief Title: Carboplatin and Paclitaxel in Treating Older Patients With Metastatic or Recurrent Unresectable Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9921; CDR0000067656 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-04-06; First posted 2004-05-26 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carboplatin + paclitaxel (Experimental): Following completion of the Lubben Social Network Scale and Frailty Questionnaire, patients receive carboplatin IV over 30 minutes and paclitaxel IV over 60 minutes on days 1, 8, and 15.
  Treatment repeats every 28 days for 2 courses. Patients with complete response receive 2 additional courses of therapy. Patients with partial response or stable disease may receive additional courses of therapy at investigator's discretion. Patients are followed every 3 months for 5 years or until disease progression.
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of carboplatin and paclitaxel in treating patients who have metastatic or recurrent unresectable non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate to carboplatin and paclitaxel in elderly patients with metastatic or recurrent unresectable non-small cell lung cancer. II. Determine the toxicity of this regimen in these patients. III. Determine if the hypothesized lack of social support impacts the recruitment of elderly patients into clinical trials. IV. Determine if a previously validated tool of functional status in the elderly predicts treatment related toxicity superior to that predicted by the ECOG performance status in this patient population.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer Stage IV disease OR Recurrent unresectable disease No other conventional curative or significant palliative therapies available Measurable disease At least one lesion a minimum of one dimension in diameter of at least 20 mm No symptomatic and/or untreated CNS metastases

PATIENT CHARACTERISTICS: Age: 65 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: AST no greater than 3 times upper limit of normal Renal: Creatinine clearance at least 40 mL/min Other: No uncontrolled infection No uncontrolled seizure disorder No uncontrolled diabetes mellitus No other malignancies within the past 3 years except adequately treated basal or squamous cell skin cancer or noninvasive carcinomas

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic or immunotherapy for recurrent or metastatic disease No concurrent biologic therapy Chemotherapy: No prior chemotherapy for recurrent or metastatic disease except as radiosensitizer No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for recurrent or metastatic disease except as adjuvant therapy At least 4 weeks since prior radiotherapy to greater than 25% of bone marrow No concurrent radiotherapy except for CNS therapy Surgery: See Disease Characteristics At least 3 weeks since prior major surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2000-01; Primary Completion 2003-07 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (18):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Ann Arbor Hematology Oncology, Ypsilanti, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Background] Jatoi A, Hillman S, Stella P, Green E, Adjei A, Nair S, Perez E, Amin B, Schild SE, Castillo R, Jett JR; North Central Cancer Treatment Group. Should elderly non-small-cell lung cancer patients be offered elderly-specific trials? Results of a pooled analysis from the North Central Cancer Treatment Group. J Clin Oncol. 2005 Dec 20;23(36):9113-9. doi: 10.1200/JCO.2005.03.7465. PMID 16361618
- [Result] Jatoi A, Hillman S, Stella PJ, Mailliard JA, Sloan J, Vanone S, Cannon MW, Kutteh L, Kanard A, Jett JR. Daily activities: exploring their spectrum and prognostic impact in older, chemotherapy-treated lung cancer patients. Support Care Cancer. 2003 Jul;11(7):460-4. doi: 10.1007/s00520-003-0449-5. Epub 2003 Mar 12. PMID 14505160
- [Result] Jatoi A, Stella PJ, Hillman S, Mailliard JA, Vanone S, Perez EA, Cannon MW, Geyer S, Wiesenfeld M, Jett JR. Weekly carboplatin and paclitaxel in elderly non-small-cell lung cancer patients (>or=65 years of age): a phase II North Central Cancer Treatment Group study. Am J Clin Oncol. 2003 Oct;26(5):441-7. doi: 10.1097/01.coc.0000027460.53907.38. PMID 14528068